CLINICAL TRIAL: NCT03702673
Title: Single-Dose, Randomized, Open-Label, 4-Period, 4-Sequence Crossover Study of Three Prototypes of K-877 CR Tablet and Two K-877 Tablets Administered to Healthy Adult Volunteers
Brief Title: Compare the Pharmacokinetic of K-877 Controlled Release (CR) and Immediate Release (IR) Tablets in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: K-877-101CR
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): K-877 CR Tablet A
  Interventions: Drug: K-877 CR Tablet A; Drug: K-877 CR Tablet B; Drug: K-877 CR Tablet E; Drug: K-877 IR Tablet
- Treatment B (Experimental): K-877 CR Tablet B
  Interventions: Drug: K-877 CR Tablet A; Drug: K-877 CR Tablet B; Drug: K-877 CR Tablet E; Drug: K-877 IR Tablet
- Treatment C (Experimental): K-877 CR Tablet E
  Interventions: Drug: K-877 CR Tablet A; Drug: K-877 CR Tablet B; Drug: K-877 CR Tablet E; Drug: K-877 IR Tablet
- Treatment D (Experimental): K-877 IR Tablet
  Interventions: Drug: K-877 CR Tablet A; Drug: K-877 CR Tablet B; Drug: K-877 CR Tablet E; Drug: K-877 IR Tablet

INTERVENTIONS:
Drug: K-877 CR Tablet A — K-877 Controlled Release Tablet A
Drug: K-877 CR Tablet B — K-877 Controlled Release Tablet B
Drug: K-877 CR Tablet E — K-877 Controlled Release Tablet E
Drug: K-877 IR Tablet — K-877 Immediate Release Tablet

SUMMARY:
A study to compare the pharmacokinetics of 3 types of K-877 controlled release tablets with a current normal K-877 tablet in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study-specific evaluation is performed.
* Subject is a healthy adult male or female aged 18 to 45 years, inclusive.
* Subject has a body mass index of 18 to 30 kg/m2, inclusive, at Screening.
* Subject meets all inclusion criteria outlined in the clinical study protocol.

Exclusion Criteria:

* Subject has clinically relevant abnormalities in the screening or check-in assessments.
* Subject has a supine blood pressure (as measured at Screening during the collection of vital signs) after resting for 5 minutes that is higher than 140 mm Hg systolic or 90 mm Hg diastolic, or lower than 90 mm Hg systolic or 60 mm Hg diastolic (males) or 50 mm Hg diastolic (females). If the initial blood pressure is out of range, blood pressure may be repeated after the subject has maintained a rested position in a quiet environment for at least 10 minutes.
* Subject has a supine pulse rate (as measured at Screening during the collection of vital signs) after resting for 5 minutes that is outside the range of 40 to 90 beats per minute. If the initial pulse rate is out of range, the pulse rate may be repeated after the subject has maintained a rested position in a quiet environment for at least 10 minutes.
* Subject does not meet any exclusion criteria outlined in the clinical study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) | Up to 24 hours after single administration
Maximum Measured Plasma Concentration (Cmax) | Up to 24 hours after single administration

SECONDARY OUTCOMES:
Treatment emergent adverse events summarized by treatment | Up to 16 days after administration

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Austin, Texas, United States